CLINICAL TRIAL: NCT01182948
Title: Comparison of Aerobic and Resistance Training Effects on Glycemic Control in Type 2 Diabetes
Brief Title: Effects of Different Types of Exercise in Type 2 Diabetes
Acronym: RAED2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Paolo Moghetti, Associate Professor of Endocrinology, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE1578
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: aerobic training; resistance training; type 2 diabetes; therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise (Experimental): The aerobic training group will use cardiovascular training devices.
  Interventions: Behavioral: Aerobic Training
- Resistance Exercise (Experimental): The resistance training group will perform exercises on weight machines and free weights.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Aerobic Training — The aerobic training group will exercise on cardiovascular training equipment. The workload will be gradually increased up to 60% of the reserve heart rate. Subjects will exercise 3 times per week for 60 min in the Fitness Centre of the Exercise and Sport Science School. Training will be carried out in small groups, under the supervision of personal trainers. During the study subjects will be instructed to follow an isocaloric diet.
  Arms: Aerobic Exercise
Behavioral: Resistance Training — The resistance training group will perform different exercises on weight machines and free weights to exercise upper and lower extremity muscles. Participants will perform 8-10 different exercises each session, alternating abdominal, upper and lower extremity exercises. Subjects will exercise 3 times per week for 60 min in the Fitness Centre of the Exercise and Sport Science School. Training will be carried out in small groups, under the supervision of personal trainers. During the study subjects will be instructed to follow an isocaloric diet.
  Arms: Resistance Exercise

SUMMARY:
The purposes of this study are: a) to compare the effects of supervised programs of aerobic training or resistance training on the metabolic control of type 2 diabetes; b) to investigate some potential pathophysiologic and molecular mechanisms underlying these effects; c) to assess whether some changes may persist over time after termination of the supervised programs.

DETAILED DESCRIPTION:
Meta-analyses of studies which evaluated the effects of interventions based upon structured exercise programs in patients with type 2 diabetes show that regular physical activity may improve glycosylated haemoglobin (HbA1c) by 0.6-0.7%. Most studies assessed the effects of aerobic exercise. However, recent data suggest that resistance training may result in similar effects. It seems likely that these beneficial results are obtained through different molecular mechanisms by aerobic training and resistance training. Consequently, these exercise modalities could be synergistic in improving the metabolic abnormalities in these subjects. On the other hand, comparison data are very limited.

Aims of the protocol are to compare the effects of aerobic training or resistance training on the metabolic control of type 2 diabetes and to investigate some potential pathophysiologic and molecular mechanisms underlying these effects.

The study will be carried out in 40 sedentary type 2 diabetic patients without diabetic complications, aged 40-70 yr, with body mass index (BMI) between 24-36 kg/m2 and HbA1c between 6.5-9.0%. Admitted diabetes treatments will be diet and oral hypoglycemic agents.

Subjects will be assigned, by a randomization schedule weighted by baseline BMI and fitness, to 2 groups of supervised exercise: aerobic training or resistance training. Training programs will have a similar volume and will be scheduled in three 60 min sessions per week for 4 months. During the study subjects will be instructed to follow an isocaloric diet. Before and at the end of the exercise training the following will be assessed: HbA1c (primary outcome), plasma glucose, lipid profile, blood pressure, insulin sensitivity (glucose clamp), body composition (Dual energy X-ray absorptiometry, DEXA), liver and muscle fat content (magnetic resonance imaging), expression in the muscle of some genes involved in ATP production, mitochondrial biogenesis and substrate utilization, markers of inflammation, oxidative stress and early vascular damage, peak oxygen uptake (VO2peak) during a maximal exercise test, other exercise tests, tissue oxygen extraction during exercise (Near-infrared spectroscopy, NIRS), energy expenditure and physical activity in daily life (metabolic Holter and questionnaire). Monitoring of blood glucose will also be carried out over a 48h period, comprising an exercise session (Continuous Glucose Monitoring System).

Metabolic features, exercise tests, body composition, daily physical activity and expression of relevant genes in the muscle will also be assessed 1 yr after completion of the training programs, to establish whether some changes may persist over time.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 24-36 kg/m2;
* HbA1c between 6.5-9.0%;
* diabetes diagnosis must have been made at least 1 yr previously;
* admitted diabetes treatments will be diet and oral hypoglycemic agents;
* baseline physical activity, estimated by the IPAQ questionnaire, lower than 1000 MET min per week;
* baseline body weight stable (changes lower than 2 kg in the last 2 months).

Exclusion Criteria:

* moderate-severe somatic or autonomic neuropathy;
* coronary heart disease;
* peripheral or cerebral vascular disease;
* preproliferative or proliferative retinopathy or chronic renal failure (serum creatinine >1.4 mg/dl in females; >1.5 mg/dl in males);
* therapy with beta-blocker drugs;
* smokers;
* acute clinically significant intercurrent diseases;
* inability to perform the scheduled physical activity programs.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in haemoglobin A1c (HbA1c) levels | 4 months
  The measurement of HbA1c is carried out with a DCCT (Diabetes Control and Complications Trial)-aligned method.

SECONDARY OUTCOMES:
Change in body weight | 4 months
Change in body composition | 4 months
  Assessment by DEXA (Dual energy X-ray absorptiometry)
Change in fasting plasma glucose levels | 4 months
Change in total cholesterol levels | 4 months
Change in HDL-cholesterol levels | 4 months
Change in LDL-cholesterol levels | 4 months
Change in triglycerides levels | 4 months
Change in blood pressure | 4 months
Change in insulin sensitivity | 4 months
  Measured by euglycemic hyperinsulinemic clamp
Change in energy expenditure | 4 months
  Measured by indirect calorimetry
Change in antidiabetic medications | 4 months
  Class and dosage of blood-glucose lowering drugs are recorded before and at the end of the protocol.
Compliance | 4 months
  Attendance at the scheduled sessions is recorded for each patient.
Change in beta-cell function | 4 months
  Measured by OGTT (Oral Glucose Tolerance Test)
Change in energy expenditure through voluntary physical activity | 4 months
  Energy expenditure is estimated through metabolic Holter (Sense Wear Armband) and IPAQ (International physical activity questionnaire).
Change in peak oxygen uptake | 4 months
  Measured during an incremental exercise test
Change in tissue oxygen extraction | 4 months
  Measured by NIRS (Near-infrared spectroscopy) during an incremental test exercise
Change in liver and muscle fat content | 4 months
  Measured by Magnetic Resonance Imaging
Change in blood glucose during and after exercise | 48 hours
  Measured by continuous glucose monitoring system
Muscle strength | 4 months
  Measured by 1RM (one-repetition maximum) test
Change in 6 minutes walk distance | 4 months
  This test measures the number of meters that can be walked in 6 minutes over a 30 m course. It is a simple field test to assess aerobic functional capacity.
Change in flexibility | 4 months
  Measured by "sit and reach" test and "back scratch" test
Changes in expression in the muscle of some genes involved in ATP production, mitochondrial biogenesis and substrate utilization | 4 months
  mRNA analysis with multiplex tandem real-time PCR of fine needle aspirates obtained from the vastus lateralis muscle

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Moghetti, MD.,Ph.D., Principal Investigator — Universita di Verona

REFERENCES:
- [Derived] Dauriz M, Olioso D, Moghetti P. Response to Comment on Olioso D, et al. "Effect of Aerobic and Resistance Training on Circulating Micro-RNA Expression Profile in Subjects with Type 2 Diabetes". J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgaa068. doi: 10.1210/clinem/dgaa068. No abstract available. PMID 32080720
- [Derived] Olioso D, Dauriz M, Bacchi E, Negri C, Santi L, Bonora E, Moghetti P. Effects of Aerobic and Resistance Training on Circulating Micro-RNA Expression Profile in Subjects With Type 2 Diabetes. J Clin Endocrinol Metab. 2019 Apr 1;104(4):1119-1130. doi: 10.1210/jc.2018-01820. PMID 30445461
- [Derived] Bellavere F, Cacciatori V, Bacchi E, Gemma ML, Raimondo D, Negri C, Thomaseth K, Muggeo M, Bonora E, Moghetti P. Effects of aerobic or resistance exercise training on cardiovascular autonomic function of subjects with type 2 diabetes: A pilot study. Nutr Metab Cardiovasc Dis. 2018 Mar;28(3):226-233. doi: 10.1016/j.numecd.2017.12.008. Epub 2018 Jan 2. PMID 29402509
- [Derived] Bacchi E, Negri C, Trombetta M, Zanolin ME, Lanza M, Bonora E, Moghetti P. Differences in the acute effects of aerobic and resistance exercise in subjects with type 2 diabetes: results from the RAED2 Randomized Trial. PLoS One. 2012;7(12):e49937. doi: 10.1371/journal.pone.0049937. Epub 2012 Dec 5. PMID 23227155
- [Derived] Bacchi E, Negri C, Zanolin ME, Milanese C, Faccioli N, Trombetta M, Zoppini G, Cevese A, Bonadonna RC, Schena F, Bonora E, Lanza M, Moghetti P. Metabolic effects of aerobic training and resistance training in type 2 diabetic subjects: a randomized controlled trial (the RAED2 study). Diabetes Care. 2012 Apr;35(4):676-82. doi: 10.2337/dc11-1655. Epub 2012 Feb 16. PMID 22344613